CLINICAL TRIAL: NCT04695275
Title: A Multicenter Observational Study About the Clinical Feature and Microbiology Characteristics of Empyema in Children
Brief Title: Clinical Feature and Microbiology Characteristics of Empyema in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); Tianjin Children's Hospital (Other); Second Hospital affiliated with Tianjin Medical University (Unknown); Children's Hospital of Hebei Province (Other); Baoding Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Director of China National Clinical Research Center for Respiratory Diseases, Chief of Respiratory Department, Beijing Children's Hospital
Other Study IDs: BCH Lung 013
Record Dates: First submitted 2020-12-14; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-03

CONDITIONS: Empyema
Keywords: Empyema; streptococcus; Children
MeSH Terms: conditions — Empyema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is designed to clarify the clinical characteristics and reversion of children with empyema, observe the effect of streptococcus vaccine application on serotype of streptococcus, and to explore the susceptibility factors of streptococcus empyema in children in China.

DETAILED DESCRIPTION:
Empyema is a major complication of bacterial community-acquired pneumonia in children. And studies have shown that although the incidence of community-acquired pneumonia in children has decreased with the application of pneumococcal conjugate vaccine, the incidence of empyema has increased, which raises the difficulty to disease treatment, and aggravates the financial burden on medical care.

Streptococcus is one of the most common pathogens causing children's empyema. In recent years, although more and more researches are reported on children's community- acquired pneumonia or pleural effusion, the clinical studies on streptococcus pneumoniae empyema are rarely mentioned. Therefore, a multicenter observational study is needed to better understand the clinical characteristics and reversion of children with empyema, observe the effect of streptococcus vaccine application on serotype of streptococcus, and explore the susceptibility factors of streptococcus empyema in children in China. The study mentioned above will contribute to optimize the treatment strategy of streptococcus empyema for the future, and reduce the incidence of children's empyema.

The trial will be completed in 3 years with 100 participants taken from hospitals in partnership with clinical research collaboration of National Clinical Research Center for Respiratory Diseases, China.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 day to 18 years
* Admitted with diagnosis of pneumonia combined with pleural effusion
* The appearance of thoracic fluid or the results of fluid examination conforms to empyema with at least 1 of the following criteria:

  * Thoracentesis is pus.
  * Thoracic fluid smear observation show bacterial-positive.
  * Thoracic fluid culture test show bacterial-positive.
  * Cell counting of thoracic fluid is more than 10x109/L.

Exclusion Criteria:

* Subjects will be excluded if the thoracic fluids are caused by non-infectious factors, such as cardiovascular, connective tissue disease, tumor or trauma, etc.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are aged 1day to 18 years, and diagnosed with "pneumonia combined with empyema"
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-06 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The cure rate of empyema | 6 months
  Percentage
The improvement rate of empyema. | 6 months
  Percentage
The incidence of long-term adverse outcomes. | 6 months
  Percentage

SECONDARY OUTCOMES:
Duration of fever | 4weeks
  Days
Duration of respiratory symptoms | 4weeks
  Days
Duration of hospitalization | 4weeks
  Days
Number of participant(s) with extra-pulmonary complications, including shock, renal failure, multiple organ failure, hemophagocytosis syndrome, et al. | 4weeks
  Number
Proportion of streptococcus pneumoniae empyema | 10 months
  Percentage
Serotype distribution of children with streptococcus pneumoniae empyema | 10 months
  Percentage
Vaccination rate of pneumococcal conjugate vaccine | 6 months
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital,, Beijing, Beijing Municipality, China